CLINICAL TRIAL: NCT06091722
Title: Quantitative Assessment of Lid Margin Vascularity Using Swept-source Optical Coherence Tomographic Angiography
Brief Title: Quantitative Assessment of Lid Margin Vascularity Using SS-OCTA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Principal Investigator, Wenzhou Medical University
Other Study IDs: 20230801LMBFD
Record Dates: First submitted 2023-10-15; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Ss-octa; Lid Margin Blood Flow Density; MGD

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Mild group, the scores of both clinicians were ≤ grade 1
- 2: Moderate group, one doctor scored grade 2, and the other doctor scored 1~2;
- 3: Moderate group, one doctor scored grade 2, and the other doctor scored 1~2;

SUMMARY:
To explore an optimized scan technique for the detection of lid margin vasculature

DETAILED DESCRIPTION:
To investigate whether the SS-OCTA tool has the potential to characterize the lid margin vascularity in MGD patients. The repeatability and validity of OCTA in assessing eyelid margin blood flow density was evaluated。

ELIGIBILITY:
Inclusion Criteria:

The MGD patients were aged >_20 years and were diagnosed according to Chinese MGD diagnostic criteria,11 including dry eye symptoms, and at least one of the following signs: (1) poor meibum expressibility or quality; (2) at least one of eyelid margin abnormalities (lid margin irregularity, plugging of the gland orifice, vascular engorgement/telangiectasia, and anterior replacement of the mucocutaneous junction. Normal subjects were defined as adults without any dry eye symptoms and lid margin abnormality.

Exclusion Criteria:

(1) subjects with ocular diseases or conditions known to affect the anatomy of the anterior segment, such as acute ocular inflammation, a history of eyelid surgery, contact lens wear within two weeks, and/or eyelid trauma; (2) subjects with of history of systemic or topical medications that might cause ocular congestion; (3) subjects with severe systemic illness or pregnancy; and (4) subjects who were difficult to cooperate with examination, resulting the obtained images were not sufficiently clear for automatic analysis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MGD or normal patients who could cooperate with dry eye evaluation and SSOCTA examination in the dry eye Clinic of the Eye Hospital of Wenzhou Medical University were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
LMBFD | Immediately after ssocta
  Lid margin blood flow density

IPD SHARING:
Plan to Share IPD: No